CLINICAL TRIAL: NCT07047014
Title: Advancing Reperfusion Therapy for Ischemic Stroke (ARTS): Tenecteplase in Medium Vessel Occlusion (MeVO) for Acute Ischemic Stroke
Acronym: ARTS-MeVO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); Chinese Stroke Association (Unknown)
Responsible Party: Principal Investigator, Yunyun Xiong, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSA2024YJ006
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-08

CONDITIONS: Stroke, Ischemic; Medium Vessel Occlusions
Keywords: ischemic stroke; tenecteplase; medium vessel occlusions; beyond 4.5 hours
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenecteplase (0.25 mg/kg) (Experimental): Tenecteplase (0.25 mg/kg, max 25 mg)
  Interventions: Drug: Tenecteplase (0.25mg/kg)
- Standard medical treatment (Active Comparator): Aspirin combined with clopidogrel, aspirin alone, or clopidogrel alone
  Interventions: Drug: Standard medical treatment

INTERVENTIONS:
Drug: Tenecteplase (0.25mg/kg) — Each vial of tenecteplase is reconstituted with 3 ml sterile water for injection and adjusted to a concentration of 5.33 mg/ml. Calculate the total amount of drug according to the subject's actual body weight and measure the required drug volume. The maximum dose should not exceed 25mg. Tenecteplase should be given as a single, intravenous bolus (within 5-10 seconds).
  Arms: Tenecteplase (0.25 mg/kg)
Drug: Standard medical treatment — Aspirin combined with clopidogrel, aspirin alone, or clopidogrel alone after randomization at the discretion of site researchers according to Chinese Guidelines for Diagnosis and Treatment of Acute Ischemic Stroke 2023.
  Arms: Standard medical treatment

SUMMARY:
Results from recent several trials provided data showing limits to the effectiveness of thrombectomy for ischemic stroke due to medium vessel occlusions.The benefit-risk profile of thrombolysis for these patients has never been investigated. We initiated a multicenter, prospective, randomized, open label, blinded-endpoint (PROBE) controlled trial to evaluate the efficacy and safety of tenecteplase (0.25mg/kg, maximum dose 25mg) compared to standard medical care for patients with acute ischemic stroke due to medium vessel occlusion (MeVO) within 4.5 to 24 hours from symptom onset.

DETAILED DESCRIPTION:
Adult acute ischemic stroke patients due to primary medium vessel occlusions (distal M2/M3 segments of the middle cerebral artery, A1/A2/A3 segments of the anterior cerebral artery, and P1/P2/P3 segments of the posterior cerebral artery confirmed by CTA/MRA, and responsible for the signs and symptoms of acute ischemic stroke) with baseline National Institutes of Health Stroke Scale (NIHSS) ≥6 or NIHSS 3-5 with disabling symptoms will be enrolled in this trial. We use perfusion imaging to select subjects and the enrolled patients have target mismatch profile on CTP or MRI+PWI (ischemic core volume <70mL, mismatch ratio>1.2, mismatch volume >10mL). We will randomly assign eligible patients to receive tenecteplase (at a dose of 0.25 mg per kilogram of body weight; maximum dose, 25 mg) or standard medical treatment 4.5 to 24 hours after the time that the patient was last known to be well (including after stroke on awakening and unwitnessed stroke). The primary outcome is the proportion of patients with an mRS score ≤ 1 at 90 days.

ELIGIBILITY:
Inclusion Criteria:

* (1)Age≥18 years old; (2)Acute ischemic stroke symptom onset within 4.5 - 24 hours; including wake-up stroke and unwitnessed stroke, onset time refers to "last-seen normal time"; (3)Primary medium vessel occlusions confirmed by CTA/MRA, including distal M2/M3 segments of the middle cerebral artery (MCA), A1/A2/A3 segments of the anterior cerebral artery (ACA), and P1/P2/P3 segments of the posterior cerebral artery (PCA) and responsible for the signs and symptoms of acute ischemic stroke; (4)Pre-stroke modified Rankin scale (mRS) score ≤1; (5)Baseline National Institutes of Health Stroke Scale (NIHSS) ≥6 or NIHSS 3-5 with disabling symptoms; (6)Neuroimaging criteria: Target mismatch profile on CT perfusion or MRI+MR perfusion (ischemic core volume <70mL, mismatch rate >1.2, mismatch volume >10mL); (7)Written informed consent from patients or their legally authorized representatives.

Exclusion Criteria:

* (1)Allergy to tenecteplase; (2)Rapidly improving symptoms at the discretion of the investigator; (3)NIHSS consciousness score 1a >2, or epileptic seizure, hemiplegia after seizures (Todd's palsy) or other neurological/mental illness such that the patient is not able to cooperate or unwilling to cooperate; (4)Intention to undergo endovascular treatment. (5)Persistent blood pressure elevation (systolic ≥185 mmHg or diastolic ≥110 mmHg), despite blood pressure-lowering treatment; (6)Blood glucose <2.8 or >22.2 mmol/L (point of care glucose testing is acceptable); (7) Active internal bleeding or at high risk of bleeding, e.g., major surgery, trauma or gastrointestinal or urinary tract hemorrhage within the previous 21 days, or arterial puncture at a non-compressible site within the previous 7 days; (8)Any known impairment in coagulation due to comorbid disease or anticoagulant use. If on warfarin, then INR >1.7 or prothrombin time >15 seconds; use of any direct thrombin inhibitors or direct factor Xa inhibitors during the last 48 hours unless reversal of dabigatran can be achieved with idarucizumab; any full dose heparin/heparinoid during the last 24 hours or with an APTT greater than the upper limit of normal; (9)Known defect of platelet function or platelet count below 100,000/mm3 (NB patients taking antiplatelet medication can be included); (10)Ischemic stroke or myocardial infarction in previous 3 months, previous intracranial hemorrhage, severe traumatic brain injury or intracranial or intraspinal operation in previous 3 months, or known intracranial neoplasm, arteriovenous malformation, or giant aneurysm; (11)Any terminal illness such that the patient would not be expected to survive more than 1 year; (12) Unable to perform CTP or PWI; (13)Hypodensity in >1/3 MCA territory on non-contrast CT or hypodensity outside the current perfusion lesion suggesting distal clot migration (secondary MeVO); (14)Acute or past intracerebral hemorrhage (ICH) identified by CT or MRI; (15)Pregnant women, nursing mothers, or reluctance to use effective contraceptive measures during the period of the trial; (16)Unlikely to adhere to the trial protocol or follow-up; (17) Participation in other interventional clinical trials within the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
mRS score ≤ 1 at 90 days | 90 days
  The proportion of patients with an mRS score ≤ 1 at 90 days

SECONDARY OUTCOMES:
mRS score | 90 days
  Ordinal distribution of mRS at 90 days (shift analysis)
mRS score ≤ 2 | 90 days
  The proportion of patients with an mRS score of 0-2 at 90 days
Early neurological improvement | 24 hours
  The rate of early neurological improvement at 24h after randomization (defined as a NIHSS score ≤1 or ≥4 points compared with the baseline)
mRS 5-6 | 90 days
  mRS 5-6 at 90 days
EuroQol 5-Dimension (EQ-5D) index | 90 days and 1 year
  EuroQol 5-Dimension (EQ-5D) index at 90 days and 1 year
mRS score at 1 year | 1 year
  mRS score at 1 year
Symptomatic intracranial hemorrhage | 36 hours
  Symptomatic intracranial hemorrhage within 36 hours (defined by the SITS-MOST criteria)
All-cause mortality | 90 days and 1 year
  All-cause mortality at 90 days and 1 year
Systemic bleeding | 90 days
  Systemic bleeding at 90 days (defined by the GUSTO criteria: moderate and severe bleeding)
Adverse events (AEs)/ serious adverse events (SAEs) | 90 days
  Adverse events (AEs)/ serious adverse events (SAEs) within 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Ziqi Xu, Principal Investigator — First Affiliated Hospital of Zhejiang University; Yunyun Xiong, Principal Investigator — Beijing Tiantan Hospital
Locations (7):
- China (7):
  - Beijing tiantan hospital, Beijing, Beijing Municipality
  - Jiuquan city people's hospital, Jiuquan, Gansu
  - Xingtang People's Hospital, Shijiazhuang, Hebei
  - Jiyuan Traditional Chinese Medicine Hospital, Jiyuan, Henan
  - The first people hospital of lingbao, Lingbao, Henan
  - Hai'an People's Hospital, Nantong, Jiangsu
  - The First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided